CLINICAL TRIAL: NCT00762814
Title: The Use of Sensory or Motor Cues Using Electrical Stimulation to Reduce Gait Freezing in Patients With Parkinson Disease
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: There was no funding for the device to be used in the study.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-0890
Record Dates: First submitted 2008-09-23; First posted 2008-09-30 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; Individuals; frequent; freezing; during; gait
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Parkinson subjects with freezing (Experimental): Each subject will have been diagnosed with Parkinson disease and will serve as his/her own control. Inclusion criteria: history of consistent freezing with ambulation in a straight line and/or when turning, normal central and peripheral neurological function, at least grade 4 strength and normal joint ranges of motion in both legs, normal somatosensory function in the feet (joint position sense), except for their neurological diagnosis and use of levodopa, each must have had clear benefit from levodopa for at least some of his/her PD symptoms, and all subjects with PD must be able to walk independently for 10 feet.
  Exclusion criteria include: serious medical problem that would impair the ability to undergo testing, use of neuroleptic or other dopamine-blocking drug, use of drugs that might affect balance, history or evidence of other neurological deficit that could interfere, such as previous stroke or muscle disease, or participants who are unable to provide informed consent.
  Interventions: Device: Gait tests with and without the use of a tactile sensory cue (electrical stimulation using a TENS unit)

INTERVENTIONS:
Device: Gait tests with and without the use of a tactile sensory cue (electrical stimulation using a TENS unit) — Eligible subjects will be perform walking tests involving the use of the TENS device (Select Unit by Empi) on the lower leg bilaterally during gait: uncued (wearing the unit but, but with the device turned off) or with a tactile cue (wearing the device with it turned on until a tactile stimulus is felt). The TENS unit is a battery-operated, single-channel electrical stimulator worn around the proximal calf that can used to provide a constant tactile stimulus. All subjects will undergo a single visit in which the two walking conditions are tested. During these visits, the patient will perform the same gait assessments measured with the device turned off as well as turned on. Testing the two conditions on the same day/time will provide the investigators with a consistent comparison of the two tested conditions, as mobility and function in patients with PD can vary significantly within and between days.

SUMMARY:
Some individuals with Parkinson disease experience "freezing" during walking which results in their inability to move their feet. They often have difficulty starting to move once they have stopped. Freezing often results in loss of balance and falling. Oral medications for Parkinson disease aren't as effective in treating freezing as it is in reducing other symptoms. Another treatment for freezing is instruction in walking using visual targets or auditory cues (thinking of a rhythm or beat). These cues can be initially effective for some individuals, but the effects do not last. Other types of cues have not been studied. We want to examine the effects of two other cues, tactile (touch) or motor (muscle contraction), on the effects of freezing.

DETAILED DESCRIPTION:
We will use a device (TENS unit) that provides electrical stimulation to a nerve in the lower legs. Electrodes will be placed on the skin of your lower legs and a box that delivers electrical current will cause a tingling feeling in the legs. Subjects will be asked to perform three gait tasks with the device on and off to compare the effects of the sensory cue on the speed/time to complete gait tasks and the frequency and duration of any freezing events. This use of the device (TENS unit) is investigational. While it has been approved by the Food and Drug Administration for the treatment of pain, it has not been approved for the treatment of freezing. Because the TENS unit can provide a sensory cue, it may help to prevent or reduce freezing. If it is found that this cue works, it could lead to new treatments for the treatment of freezing.

ELIGIBILITY:
Inclusion Criteria:

1. PD diagnostic criteria include those used for clinically defined "definite PD", as previously outlined22 based upon established criteria.22, 23
2. history of consistent freezing with ambulation in a straight line and/or when turning.
3. normal central and peripheral neurological function
4. at least grade 4 strength and normal joint ranges of motion in both legs
5. normal somatosensory function in the feet (joint position sense), except for their neurological diagnosis and use of levodopa.
6. Each must have had clear benefit from levodopa for at least some of his/her PD symptoms
7. All subjects with PD must be able to walk independently for 10 feet.

Exclusion Criteria:

1. serious medical problem that would impair the ability to undergo testing.
2. use of neuroleptic or other dopamine-blocking drug
3. use of drugs that might affect balance
4. history or evidence of other neurological deficit that could interfere, such as previous stroke or muscle disease
5. participants who are unable to provide informed consent

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-05; Primary Completion 2009-03 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go | Time of study visit

SECONDARY OUTCOMES:
Time to perform a 360 degree turn while standing in place | Time of study visit
Time to complete a figure-eight walking pattern around cones placed anterior and posterior to the subject | Time of study visit

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University Program in Physical Therapy, St Louis, Missouri, United States